CLINICAL TRIAL: NCT02716623
Title: The Feasibility of a Diet and Exercise Intervention in Diabetics During Treatment for Non-muscle Invasive Bladder Cancer
Acronym: DEAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Eugene Lee, MD, Assistant Professor, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00001802; UL1TR000001 (NIH)
Record Dates: First submitted 2016-03-10; First posted 2016-03-23 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Bladder Cancer; Diabetes Mellitus
MeSH Terms: conditions — Urinary Bladder Neoplasms; Diabetes Mellitus | interventions — Diet, Carbohydrate-Restricted; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CR Diet and Exercise (Experimental): Participants will be asked to follow specific diet intervention and exercise regimen.
  Interventions: Other: CR diet; Behavioral: Exercise

INTERVENTIONS:
Other: CR diet — Diet consists of meals lower in carbohydrates but does not restrict the number of calories that participants can consume.
  Other Names: Carbohydrate restricted diet
Behavioral: Exercise — Participants will be asked to undergo specific exercise schedule. Exercise will be tracked using a fitness device.

SUMMARY:
The purpose of this study is to learn if bladder cancer patients can follow a diet and exercise program during treatment and whether the program will improve results of their treatment.

DETAILED DESCRIPTION:
This study will examine the effects of a carbohydrate restricted (CR) diet in bladder cancer patients with diabetes. The goal of this pilot study is to determine if the CR diet and exercise routine are feasible for this patient population to follow.

Participants in this study will receive meals tailored to their specific needs. A registered dietitian will work with them to establish guidelines for the meals and to follow their progress throughout the study.

Participants will be asked to be in this study for up to 12 months. A participant will be asked to make a total of 16 in-person visits over the course of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-muscle-invasive bladder cancer
* Have completed Transurethral Resection of Bladder Tumor (TURBT) procedure
* Diagnosis of diabetes or pre-diabetes, or use diabetic medication, or show signs of diabetes which would prompt a diabetic screening

Exclusion Criteria:

* Evidence of muscle-invasion or metastatic disease
* BMI less than 18.5 and/or score in the "severe malnourished" category of the patient generated subjective global assessment (PGSGA)
* Unable to complete the exercise regimen or deemed a fall risk
* Participating in a research study involving any form of treatment intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-03; Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Participant compliance with study specific CR diet | 12 months
  Measure participant compliance with CR diet. Compliance will be measured through adherence to study diet. Study team members will regularly check in with participants to track weekly food data.

SECONDARY OUTCOMES:
Presence of Tumor M2-PK | 12 months
  Level of Tumor M2-PK will be assessed over the course the study.

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Lee, MD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas